CLINICAL TRIAL: NCT04129320
Title: A Phase 2/3 Open-Label Trial to Evaluate Enoblituzumab in Combination With MGA012 or MGD013 in the First-Line Treatment of Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Enoblituzumab Plus MGA012 or MGD013 in Squamous Cell Carcinoma of the Head and Neck
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Change in study design
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGA271-05
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Cancer; Squamous Cell Carcinoma of Head and Neck
Keywords: SCCHN; head and neck; oropharyngeal; oral cavity; hypopharyngeal; laryngeal cancer; immunotherapy; PD-1; B7-H3; LAG-3
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Laryngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel study model refers to concurrent enrollment of non-randomized Modules X and Y.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental Arm 1 (Experimental): Enoblituzumab plus MGA012
  Interventions: Biological: enoblituzumab; Biological: MGA012
- Experimental Arm 2 (Experimental): Enoblituzumab plus MGD013
  Interventions: Biological: enoblituzumab; Biological: MGD013

INTERVENTIONS:
Biological: enoblituzumab — anti-B7-H3 antibody
  Other Names: MGA271
Biological: MGA012 — anti-PD-1 antibody
  Other Names: INCMGA00012
  Arms: Experimental Arm 1
Biological: MGD013 — PD-1 X LAG-3 bispecific DART protein
  Arms: Experimental Arm 2

SUMMARY:
This is an open-label study designed to evaluate safety and efficacy of enoblituzumab in combination with MGA012 or MGD013 in first-line treatment of patients with recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN).

DETAILED DESCRIPTION:
The study will initially be conducted in 2 modules, Module X (enoblituzumab plus MGA012) and Module Y (enoblituzumab plus MGD013). Enrollment into Modules X and Y, with approximately 30 patients each, will occur independently in a non-randomized fashion. Data from these modules will determine if further evaluation will occur in randomized Module A (Phase 2) and randomized Module B (Phase 3).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven, recurrent or metastatic SCCHN not curable by local therapy
* No prior systemic therapy for SCCHN in the recurrent or metastatic setting (with the exception of systemic therapy completed > 6 months prior of given as part of multimodal treatment for locally advanced disease)
* Primary tumor locations of oropharynx, oral cavity, hypopharynx, or larynx
* At least one radiographically measurable lesion
* HPV test results available (positive and negative eligible)
* ECOG Performance status of 0 or 1
* Adequate end organ function
* Positive PD-L1 expression level (CPS ≥ 1%)

Exclusion Criteria:

* Disease suitable for local therapy administered with curative intent
* Progressive disease within 6 months of completion of curatively intended systemic treatment for locoregionally advanced SCCHN
* Radiation or other non-systemic therapy within 2 weeks of first dose of study drug
* Diagnosis of immunodeficiency, or use of immunosuppresive therapy within 14 days of first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (Modules X and Y) | 2 years
  Proportion of patients with best overall response of complete response (CR) plus partial response (PR) per RECIST 1.1
Incidence of Adverse Events as assessed by CTCAE v 4.03 (Modules X and Y) | Up to 30 days after last dose of study drug
  Evaluation of adverse events and serious adverse events

SECONDARY OUTCOMES:
Progression-free Survival - (Modules X and Y) | 2 years
  Time from start of study treatment to the first documented disease progression per RECIST v1.1 or death due to any cause, whichever occurs first.
Disease Control Rate - (Modules X and Y) | 2 years
  Percentage of patients who experienced response of CR, PR or stable disease for at least 3 months from start of study treatment
Duration of Response - (Modules X and Y) | 2 years
  Time from the date of initial response to the date of first documented progression or death from any cause, whichever occurs first
Immunogenicity (Module X) | 2 years
  Percentage of patients developing anti-drug antibodies to enoblituzumab and/or MGA012
Immunogenicity (Module Y) | 2 years
  Percentage of patients developing anti-drug antibodies to enoblituzumab and/or MGD013
Cmax (Module X) | 2 years
  Maximum serum concentration of enoblituzumab and MGA012
Ctrough (Module X) | 2 years
  Trough serum concentration of enoblituzumab and MGA012
Cmax (Module Y) | 2 years
  Maximum serum concentration of enoblituzumab and MGD013
Ctrough (Module Y) | 2 years
  Trough serum concentration of enoblituzumab and MGD013

IPD SHARING:
Plan to Share IPD: No